CLINICAL TRIAL: NCT00780676
Title: Personalized Treatment Selection for Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed early for futility.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0574; NCI-2012-01671 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-10-24; First posted 2008-10-28 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Dasatinib; Metastatic Breast Cancer; Sprycel; BMS-354825; Genetic testing; AZD6244; Selumetinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dasatinib sensitivity signature (Experimental): Participants predicted to respond to Dasatinib (Sprycel) by predictive gene signature receive dasatinib 100 mg by mouth daily.
  Interventions: Drug: Dasatinib
- SRC pathway activity signature (Experimental): Participants predicted to respond to Dasatinib (Sprycel) by predictive gene signature receive dasatinib 100 mg by mouth daily.
  Interventions: Drug: Dasatinib
- Dasatinib target index (Experimental): Participants predicted to respond to Dasatinib (Sprycel) by predictive gene signature receive dasatinib 100 mg by mouth daily.
  Interventions: Drug: Dasatinib
- Selumetinib pathway predictor (Experimental): Participants predicted to respond to selumetinib/AZD6244 by predictive gene signature (either MEK pathway activity predictor positive or MEK pathway predictor negative) receive selumetinib 75 mg by mouth twice daily (BID).
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: Dasatinib — 100 mg tablet by mouth daily
  Other Names: Sprycel; BMS-354825
  Arms: Dasatinib sensitivity signature; Dasatinib target index; SRC pathway activity signature
Drug: AZD6244 — 75 mg by mouth twice daily.
  Other Names: Selumetinib
  Arms: Selumetinib pathway predictor

SUMMARY:
The goal of this clinical research study is to learn if researchers can use genetic tests to predict who may benefit from treatment with SprycelTM (dasatinib) or selumetinib (AZD6244).

DETAILED DESCRIPTION:
The Study Drug:

Dasatinib blocks several different enzymes called protein kinases that are found in cancer cells. These enzymes are important to cancer cell growth. Blocking these kinases may stop or slow cancer growth.

AZD6244 is designed to block the growth of cancer cells by interfering with specific targeted molecules needed for tumor growth, rather than by simply interfering with rapidly dividing cells (like in traditional chemotherapy).

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take either dasatinib or AZD6244. The drug you take will be decided by your doctor based on the findings of the tumor biopsy.

* If you take dasatinib, you will take 2 dasatinib tablets by mouth once every day. The dasatinib tablets will need to be swallowed whole and can be taken with or without a meal.
* If you take AZD6244, you will take 3 tablets by mouth twice every day. The AZD6244 tablet will need to be taken with 8 ounces of water on an empty stomach (1 hour before or 2 hours after a meal) about 12 hours apart.

If you have side effects, the study doctor may decrease your dose or you may stop receiving the study drug for up to 21 days.

While you receive treatment with dasatinib or AZD6244, you may not receive other anti-cancer treatment such as chemotherapy or hormonal therapy.

If you are receiving treatment with a bisphosphonate that is given by vein (such as Aredia or Zometa), you will not be able to receive the drug during the first 8 weeks of this study. This is done in order to avoid low calcium levels in the blood. You may be able to continue to receive the study drug after the first 8 weeks.

Study Visits:

Every 4 weeks while on study, you will have a complete physical exam. Blood (about 3-4 teaspoons) will be drawn for routine tests.

* If you are taking dasatinib, at Week 4, you will have an ECG.
* If you are taking AZD6244, at Week 8, and experience heart-related side effects suggestive of cardiac problems, you will have an ECHO or multiple gated acquisition scan (MUGA).

Every 8 weeks, the scans (such as MRIs, CTs, and bone scans) and x-rays that were performed at screening will be repeated.

If you experience visual disturbances while receiving AZD6244, you will have an eye exam.

Length of Study:

You may continue taking the study drug daily for as long as you are benefitting. You will be taken off study if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

If you are taken off study because of side effects, you will have CT scans or x-rays to check the status of the disease.

This is an investigational study. Dasatinib is FDA approved to treat chronic myeloid leukemia. It is not yet FDA approved for the treatment of patients with breast cancer. At this time, the use of dasatinib in breast cancer patients is investigational. AZD6244 is not FDA approved or commercially available. Its use in this study is investigational.

The tests that will be used to find out if you can receive treatment with dasatinib or AZD6244 are also investigational.

Up to 769 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. (Turnstile One - Applies only to inclusion criteria 1 - 4): Histologically confirmed breast cancer and evidence of metastatic disease that can be biopsied with acceptable risk. Patients must agree to mandatory fine needle aspiration of the cancer for response marker determination. Patient must have a positive gene expression profile. Positive gene expression signature obtained separately on trial LAB11-0337 will also be acceptable for eligibility.
2. Patients must have measurable or evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
3. Subject, age > 18 years (the safety and efficacy of dasatinib and the appropriate dose has not been established for children).
4. Signed written informed consent including a HIPAA form according to institutional guidelines.
5. (Turnstile Two Applies Only to Inclusion Criteria 5 -17) - Therapy with Dasatinib - Patient must have a positive gene expression profile. Positive gene expression obtained separately on trial LAB11-0337 will also be acceptable for eligibility.
6. Performance status Zubrod scale 0-2 (Appendix B) within 8 days of starting therapy.
7. Full physical examination and history including documentation of weight, height, and vital signs within 8 days of starting therapy.
8. Patients may have received any number of previous therapies for metastatic breast cancer. Patients must have received, had a contraindication to, or declined treatment with an anthracycline and taxane (and Herceptin if HER-2 positive) in either the adjuvant or metastatic setting.
9. Adequate organ function assessed within 14 days of study therapy, defined as: (a)Total bilirubin </= 2.0 times the institutional Upper Limit of Normal (ULN); (b) Hepatic enzymes (AST, ALT ) </= 2.5 times the institutional ULN; (c) Serum Na, K+, Mg2+, Phosphate and Ca2+ >/= lower limit of normal (LLN); (d) Serum Creatinine < 1.5 time the institutional ULN; and (e) Hemoglobin, Neutrophil count, Platelets, PT, PTT all Grade 0-1.
10. A baseline EKG within 14 days of starting therapy, with a QTc interval not > 460 msec in women, or > 450 in men.
11. Ability to take oral medication (dasatinib must be swallowed whole).
12. Patient must agree to discontinue St. Johns Wort while receiving dasatinib therapy if previously taken.
13. Patient must agree that IV bisphosphonate therapy will be withheld for the first 8 weeks of dasatinib therapy due to risk of hypocalcemia. (After the need for Ca2+ supplementation has been assessed and levels documented to be >LLN, subjects on prior bisphosphonate may be restarted with caution at the investigator's discretion).
14. Females of childbearing potential must have a negative serum pregnancy test within 7 days of starting therapy.
15. Persons of reproductive potential must agree to use and utilize a barrier method of contraception throughout treatment and for at least 4 weeks after study drug is stopped.
16. Concurrent medications must be assessed, and patient must agree to discontinue all restricted medications within 7 days of starting therapy.
17. Stable brain metastasis for at least 3 months

Exclusion Criteria:

1. (Only turnstile II applies to Exclusion Criteria): Known allergy to study drug.
2. Concurrent medical condition which may increase the risk of toxicity, including: (a) pleural or pericardial effusion of any grade; (b) uncontrolled angina, congestive heart failure or MI within (6 months); (c) history of congenital long QT syndrome or prolonged QTc interval on pre-entry electrocardiogram > 460 msec in women and >450 msec. in men; (d) any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes); continued in excl # 3
3. Continued from exclusion # 2: (e) subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration; (f) history of significant bleeding disorder unrelated to cancer, including diagnosed congenital bleeding disorders (e.g., von Willebrand's disease) or acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies); (g) ongoing or recent (3 months) significant gastrointestinal bleeding
4. Concomitant medications with any of the following drugs should be considered for exclusion unless discontinued 7 days prior to starting dasatinib: (a) Category I drugs that prolong QT interval and are generally accepted to have a risk of causing Torsades de Pointes including: quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide, dofetilide, erythromycin, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, and domperidone. Cont. in exclusion # 5
5. Continued from exclusion criterion # 4: halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
6. CYP3A4 inhibitors. Dasatinib is primarily metabolized by the CYP3A4 enzyme. Therefore, potent inhibitors of CYP3A4 may increase dasatinib plasma concentrations: (i) ketoconazole, itraconazole, erythromycin, clarithromycin,ritonavir, atazanavir, indinavir, nefazodone, nelfinavir, saquinavir; (ii) telithromycin; and (iii) subjects should be advised not to consume substantial quantities of grapefruit juice.
7. Medications which durably inhibit platelet function or inhibit anticoagulation. Medications which directly and durably inhibit platelet function or coagulation include: (i) aspirin or aspirin-containing combinations, clopidogrel, dipyridamole, tirofiban, dipyridamole, epoprostenol, eptifibatide, cilostazol, abciximab, ticlopidine, cilostazol; and (ii) warfarin, heparin/low molecular weight heparin [e.g., danaparoid, dalteparin, tinzaparin, enoxaparin]. Exceptions: low-dose warfarin for prophylaxis to prevent catheter thrombosis, and heparin for flushes of IV lines is allowed.
8. Women who are unwilling or unable to use a barrier method of contraception to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or have a positive pregnancy test at baseline, or are pregnant or breast-feeding. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
9. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness.
10. Exclusion from Selumetinib therapy include Uncontrolled hypertension (BP >/=150/95 mmHg), Heart failure (NYHA >/= Class II), prior or current cardiomyopathy (LVEF </= 50%), Atrial fibrillation (heart rate >100 bpm), Unstable ischaemic heart disease (MI within 6 months prior, or angina requiring use of nitrates more than once weekly).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Moulder, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 10, 2009 to July 25, 2012. All recruitment performed at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 97 participants recruited, 67 were excluded from the trial before assignment to groups. No participants were assigned to "MEK Pathway Activity Predictor Positive" and "MEK Pathway Predictor Negative" Arms/Groups.
Groups:
- MEK Pathway Activity Predictor Positive: Participants predicted to respond to selumetinib/AZD6244 by predictive gene signature (MEK pathway activity predictor positive) receive selumetinib 75 mg by mouth twice daily (BID).
- MEK Pathway Predictor Negative: Participants predicted to respond to selumetinib/AZD6244 by predictive gene signature (MEK pathway predictor negative) receive selumetinib 75 mg by mouth twice daily (BID).
Period: Overall Study
Arm/Group | Dasatinib Sensitivity Signature | SRC Pathway Activity Signature | Dasatinib Target Index | MEK Pathway Activity Predictor Positive | MEK Pathway Predictor Negative
Started | 9 | 8 | 13 | 0 | 0
Completed | 9 | 8 | 13 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Individuals who were positive for more than one predictor were assigned to the marker arm for which they had the highest percentile positivity.
Groups:
- MEK Pathway Activity Predictor Positive: Participants predicted to respond to selumetinib/AZD6244 by predictive gene signature (either MEK pathway activity predictor positive or MEK pathway predictor negative) receive selumetinib 75 mg by mouth twice daily (BID).
- Total: Total of all reporting groups
Arm/Group | Dasatinib Sensitivity Signature | SRC Pathway Activity Signature | Dasatinib Target Index | MEK Pathway Activity Predictor Positive | MEK Pathway Predictor Negative | Total
Number analyzed (Participants) | 9 | 8 | 13 | 0 | 0 | 30
Age, Continuous [Median (Full Range); unit: years] | 46.5 [33 to 69] | 51.6 [36 to 60] | 54.3 [42 to 62] |  |  | 51 [33 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 13 |  |  | 30
  Male | 0 | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 13 |  |  | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit (CB) Rate (CB = Participants With Objective Tumor Response or Stable Disease > 6 Months)
Description: Rate of participants with response complete, partial response or stable disease categorized by Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. Radiological response assessments must be repeated every 8 weeks during therapy.
Time Frame: Tumor status assessed every 8 weeks during therapy, up to 6 months
Population: Selumetinib pathway predictor groups (both MEK pathway activity predictor positive and MEK pathway predictor negative) had no patients assigned to either group, and only treated participants (30) included in analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dasatinib Sensitivity Signature | SRC Pathway Activity Signature | Dasatinib Target Index
Number analyzed (Participants) | 9 | 8 | 13
Percentage of Participants | 0 | 0 | 7.7

ADVERSE EVENTS:
Time Frame: Adverse event data collected with each cycle of therapy i.e. every 28 days. Overall collection period June 2009 to July 2012.
Description: Selumetinib pathway predictor groups (both MEK pathway activity predictor positive and MEK pathway predictor negative) had no patients assigned to treatment, only treated participants (30) included in analysis and adverse event reporting. Adverse event reporting was by treatment population rather than predictive groups.
Groups:
- Dasatinib 100 mg: Participants with one of 3 predictive gene signatures (dasatinib sensitivity signature, SRC pathway activity signature and dasatinib target index) received Dasatinib 100 mg orally daily.
Arm/Group | Dasatinib 100 mg
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 100 mg (N=30)
Hematoma following biopsy (General disorders) | 1
Death (General disorders) | 2 — Unrelated
Infection, Tumor wound (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib 100 mg (N=30)
Abdominal pain (Gastrointestinal disorders) | 1
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 1
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest pain (Cardiac disorders) | 1
Chills (General disorders) | 1
Cognitive disturbance (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Constitutional Symptoms (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 13
Fever (General disorders) | 2
Gastrointestinal, Sore Mouth (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 4
Hemoglobin decreased (Blood and lymphatic system disorders) | 12
Hot flashes (Reproductive system and breast disorders) | 1
Infection, Cellulitis (Infections and infestations) | 2
Joint pain (Musculoskeletal and connective tissue disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 4
Metabolic/Laboratory (other), hyperglycemia (Metabolism and nutrition disorders) | 1
Musculoskeletal (Other) (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Nausea (Gastrointestinal disorders) | 9
Neck pain (General disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 4
Pain, Left Breast (General disorders) | 1
Pain (Other) (General disorders) | 5
Pain, Chest Wall (Cardiac disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Platelet count decreased (Blood and lymphatic system disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Serum albumin decreased (Metabolism and nutrition disorders) | 1
Serum cacium decreased (Metabolism and nutrition disorders) | 1
Serum phosphate decreased (Metabolism and nutrition disorders) | 1
Serum sodium decreased (Metabolism and nutrition disorders) | 1
Serun potassium decreased (Metabolism and nutrition disorders) | 3
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vision blurred (Eye disorders) | 2
Vomiting (Gastrointestinal disorders) | 4

LIMITATIONS AND CAVEATS:
Study terminated according to early stopping rules.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes